CLINICAL TRIAL: NCT06605222
Title: A Phase I/II, Open Label, Multicenter Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-7787 in Patients With Advanced Solid Tumors
Brief Title: A Trial of SHR-7787 Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-7787-101
Record Dates: First submitted 2024-09-14; First posted 2024-09-20 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: SHR-7787 injection monotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group: SHR-7787 injection (Experimental)
  Interventions: Drug: SHR-7787 injection

INTERVENTIONS:
Drug: SHR-7787 injection — Firstly Dose Escalation and Dose Expansion of SHR-7787 injection monotherapy should be conducted.

SUMMARY:
The study is being conducted to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of SHR-7787 injection monotherapy for patients with advanced solid tumors. To explore the reasonable dosage of SHR-7787 injection monotherapy for patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study;
2. Patients with unresectable recurrent or metastatic solid tumors;
3. There is at least one lesion could be measured;
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
5. Adequate organ functions as defined;
6. Life expectancy ≥3 months.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) metastases;
2. Subjects who had other malignancy in five years before the first dose;
3. Patients with tumor-related pain that cannot be controlled as determined;
4. Patients with serious cardiovascular and cerebrovascular diseases;
5. Uncontrollable third-space effusion, such as pleural effusion, pericardial effusion or peritoneal effusion;
6. Patients with Severe infections;
7. History of immunodeficiency;
8. History of autoimmune diseases;
9. Unresolved CTCAE Grade >1 toxicity attributed to any prior anti-tumor therapy
10. Active infection;
11. Pregnant or nursing women;
12. Known history of serious allergic reactions to the investigational product or its main ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | first dose of study medication up to 21 days
  The Maximum tolerated dose of SHR-7787 injection monotherapy
Recommended phase II dose | first dose of study medication up to 21 days
  The Recommended phase II dose of SHR-7787 injection monotherapy
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | from signature completion of ICF to 60 days after the last dose or to the beginning of the new anti-cancer therapy, whichever came first, assessed up to 24 weeks
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Incidence of Dose Limited Toxicity (DLT) | from first dose to 4 weeks
  Incidence of Dose Limited Toxicity (DLT) described in the protocol

SECONDARY OUTCOMES:
Tmax | predose, 8 h (hours), 24h, 48h, 72h, 168h post-dose
  PK parameters of single dose of SHR-7787 injection monotherapy
Cmax | predose, 8 h (hours), 24h, 48h, 72h, 168h post-dose
  PK parameters of single dose of SHR-7787 injection monotherapy
AUC0-t | predose, 8 h (hours), 24h, 48h, 72h, 168h post-dose
  PK parameters of single dose of SHR-7787 injection monotherapy
t1/2 | predose, 8 h (hours), 24h, 48h, 72h, 168h post-dose
  PK parameters of single dose of SHR-7787 injection monotherapy
ADA | 0.5 hour before first dose through study completion, an average of 1 year
  Anti-drug antibody, Immunogenicity of SHR-7787 in monotherapy
ORR | from the date of the first dose to the date of disease progression evaluated based on RECIST v1.1 criteria, death, lost to follow-up, voluntary withdrawal, or initiation of other anti-tumor treatment, whichever occurs first, assessed up to 6 months
  Objective Response Rate, Efficacy endpoints of SHR-7787 injection monotherapy in treatment of patients with advanced solid tumors

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided